CLINICAL TRIAL: NCT05517122
Title: Effect of Oral NAD+ Precursors Administration on Blood NAD+ Concentration in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2201NR
Record Dates: First submitted 2022-07-04; First posted 2022-08-26 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Healthy
MeSH Terms: interventions — Niacinamide; nicotinamide-beta-riboside; microcrystalline cellulose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Nicotinamide (NAM) (Experimental)
  Interventions: Dietary Supplement: Nicotinamide (NAM)
- Nicotinamide Riboside (NR) (Experimental)
  Interventions: Dietary Supplement: Nicotinamide Riboside (NR)
- Nicotinamide Mono Nucleotide (NMN) (Experimental)
  Interventions: Dietary Supplement: Nicotinamide Mono Nucleotide (NMN)
- Microcrystalline cellulose (Placebo Comparator)
  Interventions: Dietary Supplement: Microcrystalline cellulose

INTERVENTIONS:
Dietary Supplement: Nicotinamide (NAM) — 500 mg a day
  Arms: Nicotinamide (NAM)
Dietary Supplement: Nicotinamide Riboside (NR) — 1000 mg a day
  Arms: Nicotinamide Riboside (NR)
Dietary Supplement: Nicotinamide Mono Nucleotide (NMN) — 1000 mg a day
  Arms: Nicotinamide Mono Nucleotide (NMN)
Dietary Supplement: Microcrystalline cellulose — 500 mg a day
  Arms: Microcrystalline cellulose

SUMMARY:
Nicotinamide adenine dinucleotide (NAD) is a coenzyme playing a central role in human metabolic pathways. A recognized approach to increase NAD level is through oral supplementation of its precursors promoting NAD synthesis in vivo. NAD precursors exist in multiple forms. However, it is unclear how the various precursors compare in their ability to increase NAD levels in human blood. The purpose of this study is to compare the effect of 3 NAD precursors on whole blood NAD metabolome.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female aged 18-50 years, inclusive, at enrolment
2. Body mass index (BMI) between 18.5 to 27.0 kg/m².
3. Able to understand and to sign a written informed consent prior to study enrolment.
4. Willing and able to comply with the requirements for participation in this study.

Exclusion Criteria:

1. Known history of allergy or intolerance to the investigational products.
2. Any chronic medical condition and/or history of significant medical condition, which in the opinion of the site physician/ investigator may risk participant wellbeing/ safety, impede participant compliance with study procedures or ability to complete the study and/ or could confound the primary objectives of the study.
3. Any acute illness or any recent medical intervention including vaccination within 14 days before the first dose of investigational product.
4. Female participants who are pregnant or intending to become pregnant, lactating and/or breastfeeding. Women of childbearing potential who are not currently using medically effective forms of contraception.
5. Use of prescription drugs known to potentially interact with NAD precursors within 14 days or 5 half-lives (whichever is longer) prior to the first dose of investigational product.
6. Use of multivitamin/ multimineral supplements, NAD+ precursor supplementation (e.g., niacin, nicotinic acid or niacinamide), L-tryptophan supplementation and/ or any over-the- counter (OTC) medication promoting "healthy aging" or "anti-aging" or "longevity" up to 30 days before first dose of investigational product.
7. On a self-restricted diet, controlled diet or special therapeutic diet up to 30 days before first dose of investigational product.
8. Average alcohol consumption greater than 2 standard drinks per day over a week for males, and greater than 1 standard drink per day over a week for females. One standard drink contains 10-12 g of ethanol. Examples of standard drinks are one beer can (300 ml), one glass of wine (100 ml) or one glass of schnaps (30 ml).
9. Current smoker (e.g., cigarette, tobacco, cannabis) who exceeds 5 cigarettes per week.
10. Performing shift work or trans-meridian travel greater than two time zones within 14 days prior to the first dose of investigational product.
11. Currently participating in another research study.
12. Family or hierarchical relationships with the Clinical Innovation Lab (CIL) team.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2022-07-12 (Actual); Primary Completion 2022-11-24 (Actual); Study Completion 2022-11-24 (Actual)

PRIMARY OUTCOMES:
Determine the extent of increase in NAD+ level in whole blood, for each NAD+ precursor (NAM, NR and NMN) compared to placebo | at Day 14
  Measure the changes in whole blood NAD+ level interventions vs placebo: NAM vs placebo, NR vs placebo, NMN versus placebo by quantitative liquid chromatography-mass spectroscopy
Compare the extent of increase in NAD+ level in whole blood across the 3 NAD+ precursors (NAM, NR and NMN) | at Day 14
  Measure the changes in whole blood NAD+ level across interventions: NAM vs NR, NAM vs NMN, NR vs NMN by quantitative liquid chromatography-mass spectroscopy

SECONDARY OUTCOMES:
Determine the extent the NAD+ precursors(NAM, NR and NMN) affect the NAD metabolome in whole blood compared to placebo | over 4 hours at Day 1 and at Day 14.
  Measure the change in whole blood NAD+ metabolites iAUC (reported as microM*h) and Cmax (microM) by quantitative liquid chromatography-mass spectroscopy
Compare the extent the NAD+ precursors (NAM, NR and NMN) affect the NAD+ metabolome in whole blood. | over 4 hours at Day 1 and at Day 14.
  Measure the change in whole blood NAD+ metabolites iAUC (reported as microM*h) and Cmax (microM) determined by quantitative liquid chromatography-mass spectroscopy

OTHER OUTCOMES:
Comparer the extend the NAD+ precursors (NAM, NR and NMN) affect the NAD+ metabolome in in plasma. | over 4 hours at Day 1 and at Day 14.
  Measure the change in plasma NAD+ metabolites iAUC (reported in microM) and Cmax (microM) determined by quantitative liquid chromatography-mass spectroscopy
Comparer the extend the NAD+ precursors (NAM, NR and NMN) affect the NAD+ metabolome in urine | at baseline Day 14 versus Day 1
  Measure the change in urine NAD+ metabolites iAUC (reported in microM) and Cmax (microM) determined by quantitative liquid chromatography-mass spectroscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Nestlé Clinical Innovation Lab, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Christen S, Redeuil K, Goulet L, Giner MP, Breton I, Rota R, Frezal A, Nazari A, Van den Abbeele P, Godin JP, Nutten S, Cuenoud B. The differential impact of three different NAD+ boosters on circulatory NAD and microbial metabolism in humans. Nat Metab. 2026 Jan 15. doi: 10.1038/s42255-025-01421-8. Online ahead of print. PMID 41540253